CLINICAL TRIAL: NCT00407654
Title: Phase II Trial of VEGF Trap in Patients With Previously Treated Metastatic Colorectal Cancer
Brief Title: VEGF Trap in Treating Patients With Previously Treated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00176; PHL-050 (Other Grant/Funding Number: N01CM62203); CDR0000518293 (Other Grant/Funding Number: N01CM62203); N01CM62203 (NIH)
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Results first posted 2015-08-18 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive VEGF Trap (aflibercept) IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: aflibercept

INTERVENTIONS:
Drug: aflibercept — Given intravenously
  Other Names: vascular endothelial growth factor trap; VEGF Trap; Zaltrap; ziv-aflibercept

SUMMARY:
This phase II trial is studying how well VEGF Trap works in treating patients with previously treated metastatic colorectal cancer. VEGF Trap may stop the growth of colorectal cancer by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate (complete and partial) in patients with previously treated metastatic colorectal cancer treated with VEGF Trap.

II. Determine the incidence of disease stabilization, in terms of 4-month progression-free survival, in patients treated with this drug.

SECONDARY OBJECTIVES:

I. Determine the median survival time of patients treated with this drug. II. Determine the 1-year survival rate and stable disease rate in patients treated with this drug.

III. Determine the response or stable disease duration in patients treated with this drug.

IV. Determine the toxicity of this drug in these patients. V. Determine the time to disease progression in patients treated with this drug.

VI. Determine if changes in free VEGF Trap levels correlate with response or toxicity.

OUTLINE: This is a multicenter, open-label study.

Patients are stratified according to prior bevacizumab treatment (yes vs no). Patients receive VEGF Trap IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood collection at the beginning of each course and at 60 days after completion of study treatment. Samples are analyzed by immunoenzyme techniques to determine the pharmacokinetics of VEGF Trap.

After completion of study treatment, patients are followed at 30 and 60 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* histologically/cytologically confirmed metastatic colorectal metastatic cancer
* measurable disease (at least 1 lesion accurately measured in at least 1 dimension (longest diameter) as>20mm with conventional techniques or as >10mm with spiral CT scan
* >=4 weeks from major surgery
* at least 1prior line of systemic therapy for metastatic disease. Prior treatment with anti-epidermal growth factor receptor inhibitors is allowed. Last dose >=4 weeks prior to randomization
* Two cohorts: 1) bevacizumab naïveand; 2) bevacizumab treated
* May have received prior thymidylate synthetase inhibitor concurrently with radiation as "radiation sensitizer". Last dose >=4 weeks prior to randomization
* Prior radiation treatment >=4 weeks prior to randomization
* Age>=18 years
* Life expectancy >=3 months
* ECOG<=2 (Karnofsky=60%)
* leukocytes >3.0x10^9/L
* absolute neutrophil count >1.5 x 10^9/L
* platelets>75x10^9/L
* INR <1.5 unless on warfarin
* total bilirubin within 1.5xULN
* AST/ALT≤2.5 X institution ULN
* creatinine≤1.5xULN OR creatinine clearance >60mL/min/1.73m2 for patients with creatinine levels above1.5x institution limits
* Urinalysis negative for protein OR 24h urine for protein <500 mg
* full-dose anticoagulants with PT INR >1.5 eligible provided that: a) patient is therapeutic on stable dose of warfarin or low molecular weight heparin; b) patients on warfarin, the upper target for INR is <=3; c) no active bleeding/pathological condition carrying high bleeding risk
* Eligibility of patients receiving medications known to affect activity/PK of VEGF Trap will be determined by PI
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 6 months after completion of VEGF Trap therapy
* Ability to understand/willingness to sign written informed consent

Exclusion Criteria:

* chemotherapy/radiotherapy within 4 weeks (6 weeks for nitrosoureas/mitomycin C) prior to study entry
* Other investigational agents concurrently
* History of prior anti-angiogenic therapy other than bevacizumab
* Evidence of CNS disease
* Known hypersensitivity to Chinese hamster ovary cell products/other recombinant human antibodies, and patients with a history of allergic reactions attributed to compounds of similar chemical/biologic composition to other agents used in the study.
* Serious/non-healing wound/ulcer/bone fracture
* History of abdominal fistula/GI perforation/bowel obstruction/intraabdominal abscess within 28 days of treatment
* major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 therapy
* anticipation of need for major surgical procedures during study
* core biopsy within 7 days prior to Day 1 therapy
* Patients with clinically significant cardiovascular disease
* Evidence of bleeding diathesis or coagulopathy
* PT INR >1.5 unless the patient is on full-dose warfarin
* Use of thrombolytic agents within 1 month of study initiation
* Significant Proteinuria (>500mg/24h): Urine protein should be screened by random urinalysis for protein. If dipstick positive (>1+), 24-hour urine protein should be obtained and if >500mg/24 h, patient will be excluded.
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection or psychiatric illness/social situations that would limit compliance with study
* Pregnant women
* HIV-positive patients on combination antiretroviral therapy are ineligible because of potential for PK interactions with VEGF Trap

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Moore, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (1):
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- VEGF Trap IV Arm I: Patients receive VEGF Trap IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  ziv-aflibercept: Given intravenously
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Period: Overall Study
Arm/Group | VEGF Trap IV Arm I
Started | 75
Completed | 75
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Patients receive VEGF Trap IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  ziv-aflibercept: Given orally
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Arm/Group | Arm I
Number analyzed (Participants) | 75
Age, Continuous [Median (Full Range); unit: years] | 59 [39 to 80]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 46
Region of Enrollment [Number; unit: participants]
  Canada | 49
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response (Defined as Partial or Complete Response as Defined by the RECIST Criteria)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions:Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: Up to 6 years
Measure: Number; unit: participants
Groups:
- Arm I: Patients receive VEGF Trap IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  ziv-aflibercept: Given intravenously
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Arm/Group | Arm I
Number analyzed (Participants) | 75
participants | 1

2. Primary Outcome: Progression-free Survival (Bevacizumab- naïve Group)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
  Kaplan-Meier method will be used.Progression-free survival (Bevacizumab- naïve group)
Time Frame: 4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 24
months | 2.0 [1.7 to 8.6]

3. Primary Outcome: Progression-free Survival (Bevacizumab-treated Group)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
  Kaplan-Meier method will be used. Progression-free survival (Bevacizumab-treated group)
Time Frame: 4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 51
months | 2.4 [1.9 to 3.7]

4. Secondary Outcome: Overall Survival (Bevacizumab-naïve Group)
Description: Kaplan-Meier method will be used. (Bevacizumab- naïve Group)
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 24
months | 10.4 [7.6 to 15.5]

5. Secondary Outcome: Overall Survival (Prior Bevacizumab Treated Group)
Description: Kaplan-Meier method will be used (Bevacizumab-naïve Group)
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 50
months | 8.5 [6.2 to 10.6]

6. Secondary Outcome: Time to Progression
Description: Kaplan-Meier method will be used.
Time Frame: 12 months
Population: data were not collected
Arm/Group | Arm I
Number analyzed (Participants) | 0

7. Secondary Outcome: Objective Stable Disease Rate
Time Frame: Up to 6 years
Population: data were not collected
Arm/Group | Arm I
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Response (Bevacizumab-naïve Group)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions; Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD;
  Stable disease for atleast 16 weeks
Time Frame: Up to 6 years
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 24
participants | 5

9. Secondary Outcome: Overall Survival (Bevacizumab-treated Group)
Description: Kaplan-Meier method will be used. (Bevacizumab-treated Group)
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 51
months | 8.5 [6.2 to 10.6]

10. Secondary Outcome: Overall Survival (Bevacizumab-treated Group)
Description: Kaplan-Meier method will be used (Bevacizumab-treated Group)
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 51
months | 8.5 [6.2 to 10.6]

11. Secondary Outcome: Number of Participants With Response (Bevacizumab-treated Group)
Description: as for outcome 8
Time Frame: Up to 6 years
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 50
participants | 6

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 19/75
Other Adverse Events (participants affected / at risk) | 75/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=75)
Aspartate aminotransferase increased (Investigations) | 1
Rectal pain (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Hypertension (Vascular disorders) | 2
Weight loss (General disorders) | 1
Pain (General disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
DeathNOS (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Chest pain - cardiac (Cardiac disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1
Extrapyramidal disorder (Nervous system disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=75)
Fatigue (General disorders) | 65
Hypertension (Vascular disorders) | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less